CLINICAL TRIAL: NCT02470143
Title: Pilot Study, How a Bike Application Can Support Cardiac Patients in Their Rehabilitation Program?
Brief Title: a Bike Application to Support Cardiac Patient
Acronym: BackonBike
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, prof. dr. Paul Dendale, prof. dr., Hasselt University
Other Study IDs: PDEN-IFRE 02
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Coronary Artery Disease
Keywords: Human-computer interaction; Fear; Motivation; Usability
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bike application arm: The bike application arm contains cardiac patients that will be instructed to use the cycling application during a one month period.
  Interventions: Behavioral: Bike application arm

INTERVENTIONS:
Behavioral: Bike application arm — The intervention patients will use the cycling application on a smartphone, in combination with a wrist-worn heart rate monitor. During the study, the patients will use the cycling application for one month, in which they can make use of the cycling application each time they are cycling outdoor in their home environment.

SUMMARY:
The pilot study will investigate the usability of a mobile cycling application in a cardiac patient population during a one month study period.

The application's effectiveness regarding ability to reduce fear and increase motivation to exercise will be assessed.

DETAILED DESCRIPTION:
This pilot study investigates the use of a mobile cycling application for patients with a cardiac disease that was developed by the Expertise Centre for Digital Media of Hasselt University in collaboration with the Faculty of Medicine & Life Sciences of Hasselt University. During the pilot study, the use of the cycling application and its impact on fear and motivation of patients with a cardiac disease during the rehabilitation is studied. The cycling application will be used on a smartphone, in combination with a wrist-worn heart rate monitor.

During the study, the patients will use the cycling application for one month, in which they can make use of the cycling application each time they are cycling outdoor in their home environment. Through questionnaires and interviews, the patients' experiences with respect to fear and motivation will be collected. Furthermore, the usability of the cycling application is evaluated through these questionnaires and interviews.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease for which they received a percutaneous coronary intervention, coronary artery bypass grafting or drugs only.
* Patients that have completed the standard cardiac rehabilitation program
* Patients who have access to a computer and a WiFi internet connection
* Patients that are able to go to the rehabilitation centre ReGo of Jessa Hospital
* Patients who signed the informed consent document

Exclusion Criteria:

* Patients with a history of VF, sustained VT and/or supraventricular tachycardia during the last 6 months before enrollment.
* Patients who due to cognitive, neurological and/or musculoskeletal constraints are unable to ride a bicycle.
* Patients with a pacemaker.
* Non-Dutch speaking patients
* Patients who simultaneously participate in another study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Low risk coronary artery disease patients that completed phase II of cardiac rehabilitation.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2015-08; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Impact on motivation | up to week 4

SECONDARY OUTCOMES:
Usability of the cycling application | Up to week 4
  By means of a questionnaire and an interview, the participants are asked about the usability of the application. This information will give insights in parts of the application that could be improved considering the usability.
Impact on fear | up to week 4
  By means of a questionnaire and an interview, questions are asked about participants' motivation for a tour

CONTACTS AND LOCATIONS:
Overall Officials: Ines Frederix, drs., Study Chair — Universiteit Hasselt/ Jessa ziekenhuis
Locations (1):
- Jessa Ziekenhuis, Hasselt, Belgium